CLINICAL TRIAL: NCT04310033
Title: Impact of ICU on the Quality of Life and Oncological Care of Patients With Solid Tumors
Brief Title: Impact of ICU on the Quality of Life in Cancer Patients
Acronym: QdV-ONCOREA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.420; 2019-A03307-40 (Other: ID RCB)
Record Dates: First submitted 2020-02-20; First posted 2020-03-17 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Solid Tumor, Adult
Keywords: Quality of life; Oncological care; intensive care unit; solid tumor
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: * > 18 years old
  * Non-opposition of the patient or relatives
  * Lung, head and neck or colorectal cancer
  * Non scheduled ICU admission
  * At least 24 hours of ICU stay
  * Alive at ICU discharge
  * Able to answer by phone to quality of life questionary
  Interventions: Other: Questionnaires
- Controls: Cancer patients not admitted in ICU, matched with the cases according to
  * the type of primary cancer
  * the presence or absence of oncogenic addiction
  * the setting of anticancer treatment (curative/palliative)
  * the line of anticancer treatment (none/L1/L2-L3/>L3).
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Quality of life questionary: 36-Item Short Form Survey Instrument (36-SF) at 3 and 6 months from inclusion By phone

SUMMARY:
This is an observational, prospective, monocentric, case-control study. Investigators aim to compare the quality of life and oncological treatment strategy in cancer patients admitted or not in ICU.

DETAILED DESCRIPTION:
Inclusion of cancer patients (cases) at discharge of surgical, cardiovascular and thoracic and medical ICU of the Grenoble Alpes University Hospital.

Cases will be matched with cancer patients identified in oncologist's consultation.

Inclusion of controls from oncologist consultations (2 controls for 1 case) For cases and controls, medical data will be collected at inclusion, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* > 18 ans
* Non-opposition of the patient or relatives
* Lung, head and neck or colorectal cancer
* Non scheduled ICU admission
* At least 24 hours of ICU stay
* Alive at ICU discharge
* Able to answer by phone to quality of life questionary

Exclusion Criteria:

* Unable to answer by phone to quality of life questionary
* Patient participating in another clinical study that could interfere with the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung, head and neck or colorectal cancer admitted in ICU (cases) or not (controls)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
quality of life questionary 36-item short form survey instrument (36-SF) | 3 months
  score of 0 (poor quality of life) to 100 (very good quality of life)

SECONDARY OUTCOMES:
intensity of antitumoral treatment compared to standard treatment | 3 months
  standard treatment vs adaptated treatment vs palliative care standard treatment was defined by the treatment recommended in the ESMO guidelines for each cancer (lung, colorectal, and head and neck cancer)
quality of life questionary 36-item short form survey instrument (36-SF) | 6 months
  score of 0 (poor quality of life) to 100 (very good quality of life)
intensity of antitumoral treatment compared to standard treatment | 6 months
  standard treatment vs adaptated treatment vs palliative care standard treatment was defined by the treatment recommended in the ESMO guidelines for each cancer (lung, colorectal, and head and neck cancer)
ECOG - Performance status | 3 months and 6 months
  From 0 (fully active) to 5 (dead)
Activities of Daily Living | 6 months
  From 0 (dependent ) to 6 (autonomous)
Hospital Anxiety and Depression Scale | 3 months and 6 months
  Anxiety scale from 0 (no anxiety) to 21 (anxiety) Depression Scale from 0 (no depression) to 21 (depression)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, Grenoble, France